CLINICAL TRIAL: NCT04805255
Title: Hypofractionated Stereotactic Radiotherapy for Treating Brain Oligometastases - A Prospective Longitudinal Neurocognitive Study
Brief Title: A Neurocognitive Study in Patients With Brain Oligometastases Receiving Hypofractionated SRT
Acronym: HF-SRT
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002369A3
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Brain Metastases, Adult
Keywords: Brain Oligometastases; Stereotactic Radiotherapy (SRT); Hypofractionation; Hypofractionated Stereotactic Radiotherapy (HF-SRT); Neurocognitive Functions (NCFs); Time to Progression (TTP); Time to CNS Progression; Progression-free Survival (PFS); Hippocampus; CNS Patterns of Failure; Radiation Necrosis
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypofractionated Stereotactic Radiotherapy (HF-SRT): A prospective cohort study addressing both neurocognitive outcome measures and oncological endpoints will be carried out for treating newly-diagnosed brain oligometastases with a pre-defined course of hypofractionated stereotactic radiotherapy (HF-SRT) in cancer patients with a fair/satisfactory performance status.
  Either a limited number of brain metastases or oligometastatic brain disease refers to that the number of brain metastatic lesions (both post-resected and intact) at enrollment should be limited to three or fewer and that the greatest diameter of any metastatic lesion (either a tumor bed post-surgical resection or an intact brain metastasis) should be no more than 4 cm.
  Interventions: Radiation: Hypofractionated Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiotherapy — A course of hypofractionated stereotactic radiotherapy (HF-SRT) is delivered within 2 weeks with a cumulative dose of 3000 - 3500 cGy in 5 fractions.

SUMMARY:
Background:

For newly-diagnosed patients with brain metastasis, conventional whole-brain radiation therapy (WBRT) might still remain a common palliative management even for those with brain oligometastases. However, WBRT-related late consequences, particularly a decline in neurocognitive functions (NCFs), are a major concern. Actually, WBRT-related neurocognitive dysfunction is usually characterized as deterioration involving learning and memory, in which the extremely radiosensitive hippocampus indeed plays a critical role. In order to postpone or mitigate the effect of conventional WBRT-induced neurocognitive impairments, there have been some strategies and options in clinical practice. Among them, the technique of highly precise and accurate stereotactic radiosurgery or stereotactic radiotherapy (i.e., hypofractionated stereotactic radiotherapy, HS-SRT) might have been widely administered in irradiating purely focal metastatic foci in cancer patients with a limited number of brain metastases.

Methods:

Newly-diagnosed cancer patients harboring 1-3 brain metastatic lesions are eligible if they are still in a fair/good performance status. All recruited patients should receive baseline brain MRI examination and pre-radiotherapy neurocognitive assessment. Sticking to the principles of stereotactic radiosurgery/radiotherapy (SRS/SRT), treatment planning will be designed via the technique of volumetric-modulated arc therapy (VMAT) to achieve both satisfactory in-field local control (but assuring of hippocampal avoidance) and a tolerably low incidence of radiation necrosis, a course of hypofractionated stereotactic radiotherapy (HF-SRT) is delivered within 2 weeks with a cumulative dose of 3000 - 3500 cGy in 5 fractions. Accordingly, a battery of neuropsychological measures, which includes 7 standardized neuropsychological tests (e.g., executive functions, verbal and non-verbal memory, working memory, and psychomotor speed), is used to evaluate neurocognitive functions for our registered patients. The primary outcome measure is cognitive-deterioration-free survival, which is defined mainly as the time from enrollment to a NCF decline of exceeding than 1 SD away from the baseline involving at least one of the assessed NCF tests. Additionally, patients who expire before 6 months or are alive but fail to undergo all the neurocognitive testing administered would also be defined as suffering from cognitive deterioration. There are quite a few secondary endpoints of interest, including the patterns of (CNS) failure, actual local control rates, time to (CNS) progression, and cumulative incidence of radiation necrosis.

Expected results:

This prospective neurocognitive study aims to examine thoroughly the impact of the technique of highly focal brain irradiation administered with a course of hypofractionated SRT delivered to brain metastatic lesions merely (but sparing hippocampal structures), on neurocognitive performance, time to (CNS) progression, and patterns of (CNS) failure, in patients with brain oligometastases and a fair/good performance status. It is anticipated that (in-field) local control would be durable and that neurocognitive outcomes would also be maintained favorably. Moreover, we also expect that the patterns of (CNS) failure and the individual time to progression will be clearly demonstrated in this prospective longitudinal neurocognitive study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically-confirmed non-hematopoietic malignancy who are referred for postoperative adjuvant or therapeutic hypofractionated stereotactic radiotherapy (HF-SRT).
* A Fair/good performance status no worse than Eastern Cooperative Group (ECOG) of 2 or an acceptable performance status of Karnofsky Score (KPS) at least 70.
* The number and extent of brain metastatic lesions should be no more than three metastatic foci with a greatest diameter no more than 4 cm shown on pre-radiotherapy MRI; namely, that is the clinical setting of oligometastatic brain disease or brain oligometastases.

Exclusion Criteria:

* Patients with their primary cancer arising from hematological malignancies (i.e., malignant lymphomas, leukemia), germ cell tumors, or malignant meningiomas
* Patients with MRI-identified metastasis within 5 mm peri-hippocampally
* Patients with metastasis involving the brain stem
* Clinical suspicion of leptomeningeal spreading
* History of prior radiotherapy including stereotactic radiosurgery delivered to brain/head region for any reasons

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly-diagnosed brain oligometastases and an acceptable performance status would receive baseline neurocognitive assessment.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
The cognitive-deterioration-free survival | from baseline up to 24 months
  The time from enrollment to a decline of exceeding than 1SD away from the baseline in at least one of the assessed NCF tests. Furthermore, regarding cognitive-deterioration-free survival, patients who expire before 6 months or are alive but do not undergo all the neurocognitive testing administered or even fail to receive MMSE evaluation would be assumed reasonably that they suffer cognitive deterioration at the time of death or at the time point, or they fail to receive their first neurocognitive assessment follow-up as long as there are no subsequent NCF assessments.

SECONDARY OUTCOMES:
Overall survival (OS) or Median survival time (MST) | up to 24 months
Patterns of CNS failure | up to 24 months
  1. In-field (brain) local recurrence:
     Local surgical bed recurrence Local recurrence of unresected metastases (The individual time to event is the time from study enrollment to recurrence at the local surgical bed, and the time from enrollment to progression of intact metastases, respectively.)
  2. Distant (brain) parenchymal progression
  3. Development of leptomeningeal disease (LMD)
Time to progression (TTP) | up to 24 months
Progression-free survival (PFS) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan